CLINICAL TRIAL: NCT00701480
Title: Randomized Double-Blind Case Control Study of Safety and Efficacy of Skin Cleanser Contained Hibiscus Sabdariffa Extract in Acne Treatment.
Brief Title: Safety and Efficacy of Skin Cleanser Contained Roselle Extract in Acne
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thammasat University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Mali Achariyakul/Dr., Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MTU-E-1-002/51
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2008-06-19 (Estimated); Status verified 2008-06

CONDITIONS: Acne
Keywords: acne; skin cleanser; Hibiscus sabdariffa; Roselle; safety; efficacy
MeSH Terms: conditions — Acne Vulgaris | interventions — Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): skin cleanser contained Hibiscus sabdariffa
  Interventions: Other: skin cleanser contained Hibiscus sabdariffa extract
- 2 (Active Comparator): marketed skin cleanser
  Interventions: Other: marketed skin cleanser

INTERVENTIONS:
Other: skin cleanser contained Hibiscus sabdariffa extract — face washing 2-3 times/day
  Other Names: Roselle skin cleanser
  Arms: 1
Other: marketed skin cleanser — face washing 2-3 times/day
  Other Names: Clean and Clear; Clearasil; Neutrogena
  Arms: 2

SUMMARY:
Skin cleanser for daily used is essential and one of the most common questions asked by acne patients. There are studies reported beneficial effects of cleansers in acne treatment. Extracts of plants as active ingredients in skin cleansers are increasingly popular worldwide. Roselle is a common tropical shrub. Usually, the calyces of the plant have been used to make beverages but it also used in Thai traditional medicine for several purposes including as antiseptic and astringent. The extract of roselle showed antioxidant and keratolytic effects from previous studies which fit to the pathogenesis of acne. The aims of the study is to determine the safety and efficacy of skin cleanser contained roselle extract in acne.

DETAILED DESCRIPTION:
Acne is one of the most common skin problems in teenagers and adolescents. Keys pathogenesis of the disease are 1.abnormal hypercornification of pilosebaceous duct,2.excess sebum production, 3.inflammation, 4.the present of Propionibacterium acnes. Treatments often include combination of topical and oral medications according to degree of acne severities. Acne medications can lead to drying and irritation of skin. Proper skin cleansing is important and can improve tolerability and efficacy of acne treatment.

Traditional medicine with longstanding used of herbal ingredients for skin problems and beauty is increasing more popular. Hibiscus sabdariffa L.(Roselle) is used as food, drink and topical formulation for skin infection in Thai traditional medicine. The extract from calyces contained polyphenolic compounds and anthocyanins that showed antioxidant and keratolytic activities. There for skin cleanser with Roselle extract might be benefit to acne by loosen comedone, reduce Propionibacterium acne and prevent keratinocyte injury.

The purposes of this study is to evaluate skin cleanser contained Roselle extract in two aspects ; 1. safety for irritation and allergic effects, 2. efficacy in acne as cleanser alone and as supportive care with others acne therapies.

ELIGIBILITY:
Inclusion Criteria:

* age 12-45 yrs,both sex
* clinical diagnosis of mild to moderately severe acne vulgaris(grade 1-3)
* have at least 10 facial acne lesions
* not changing any acne treatment during study period
* able to follow up according to protocol
* Written informed consent

Exclusion Criteria:

* pregnant or breast feeding
* severe acne(grade4 or nodulocystic acne)
* treated with isotretinoin orally during the last 3 months
* have other systemic disease or illness
* have allergic history to Roselle

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-07 (Estimated); Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
1. Safety evaluation: Patch test 2. Efficacy evaluation: Acne lesions counts/ acne severity grading | 6 weeks

SECONDARY OUTCOMES:
1. Safety evaluation: "a." Skin properties by visual and tactile features., "b." Biophysical parameters of skin. 2.Efficacy evaluation: Patient assessments. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mali - Achariyakul, MD., Principal Investigator — Thammasat University
Locations (1):
- Thammasat University, KlongLaung, Pathumtanee, Thailand